CLINICAL TRIAL: NCT02847195
Title: Evaluation of Pupillometry to Assess Analgesia in Children Unable to Communicate Verbally in Pediatric Intensive Care Unit (PICU)
Brief Title: Pupillometry in Pediatric Intensive Care Unit (PICU)
Acronym: Pupillomètre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL15_0642; 2013-A01600-45 (Other: ID-RCB)
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Pediatric Intensive Care
Keywords: pediatric intensive care; pain assessment; tracheal aspiration; sedation; pupillometer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pediatric intensive care (Experimental): When aspiration is planned, pain assessment will be performed thrice :
  3-5 minutes before aspiration, during aspiration, and 3-5 minutes after aspiration.
  Pain assessment will be performed with both methods:
  * COMFORT B scale (routinely performed by nurses, and lasts less than one minute)
  * Simultaneously pupillometry is assessed using the device (Neurolight) (one measurement per eye, this also lasts less than one minute) These measurements can occur at any time during stay in ICU, and can be repeated.
  Interventions: Device: pupillometry

INTERVENTIONS:
Device: pupillometry — This is a safe and painless examination (the device is simply placed on the orbit of the eye). The optical pupillometer is cleaned by doctors before and after each use, using cleaning wipes containing antibacterial, antiviral and antifungal drugs; such wipes are already in use in the service for cleaning equipment.

SUMMARY:
Assess the depth of sedation and analgesia in pediatric intensive care is critical to the management of intubated patients under mechanical ventilation. The responsiveness of the pupil is changed by the sedation and analgesia. Measuring the pupil diameter is proposed in anesthesia and intensive care to assess the quality of analgesia in adult population. Visually measuring the diameter of the pupil remains very imprecise, but this measure can be accurately and quickly performed thanks to portable devices called Pupillometers. Some devices including Algiscan® device (IdMed ) can measure in addition to the pupil diameter, the variation of pupil diameter, the latency of the pupillary reflex and the maximum speed of contraction. Pupillometry was tested in adult ICU patients, during painful and painless procedures [1]. In this study, pupillometry was more sensitive for detecting pain compared to the change in heart rate or bispectral index. The objective of this work is to perform measurements of pupil diameter during painful procedures (e.g. tracheal aspiration) in PICU. In parallel we will continue using the Comfort B-scale (has been validated for assessment of pain in children admitted to a pediatric intensive care unit [2-5] and compare the results of both types of assessment pain.

ELIGIBILITY:
Inclusion Criteria:

* children (age < 18 years) hospitalized in PICU
* sedated because they are receiving mechanical ventilation,
* for whom parents (or their representatives) have given their oral consent after written information.

Exclusion Criteria:

* children receiving curare drugs
* with congenital or acquired neurological,
* with ophthalmologic pathology
* or who does not benefit from social insurance coverage.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
pupillary diameter | Day 1
  Estimate the performances of the variation of the pupillary diameter to assess pain in children admitted in PICU in comparison to results from the COMFORT-B scale taken as reference.
  Pupillometry is assessed using a specific device the Neurolight™ (ID MED™, France), (diagnostic test under evaluation), and compared to pain assessment using the score Comfort B scale ( hetero score assessment of pain in children sedated routinely used in PICU to evaluate pain).
Comfort B Score | Day 1
  Estimate the performances of the variation of the pupillary diameter to assess pain in children admitted in PICU in comparison to results from the COMFORT-B scale taken as reference.
  Pupillometry is assessed using a specific device the Neurolight™ (ID MED™, France), (diagnostic test under evaluation), and compared to pain assessment using the score Comfort B scale ( hetero score assessment of pain in children sedated routinely used in PICU to evaluate pain).

SECONDARY OUTCOMES:
Latency time | Day 1
  Latency time assessed by the video pupillometer
pupil diameter variation | Day 1
  Pupil diameter variation assessed by the video pupillometer
diameter variation time | Day 1
  Diameter variation time assessed by the video pupillometer

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne BORDET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- service de réanimation pédiatrique, Hôpital Femme Mère Enfant (HFME), Hospices Civils de Lyon, 59 Boulevard Pinel, Bron, France